CLINICAL TRIAL: NCT02797756
Title: Impact of Gastroesophageal Reflux and Aspiration on Airway Inflammation and Microbiome in Children With Chronic Cough
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01021
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Chronic Cough (CC); Gastroesophageal Reflux (GER)
MeSH Terms: conditions — Chronic Cough; Gastroesophageal Reflux | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Case: CC/GER+ presence of chronic cough and presence of GER evidenced by esophago-gastro-duodenoscopy (EGD) with biopsy and Esophageal Impedance Monitoring (EIM) Control: CC/GER- presence of chronic cough and absence of GER by esophago-gastro-duodenoscopy (EGD) with biopsy and Esophageal Impedance Monitoring (EIM)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: CC/GER+ presence of chronic cough and presence of GER evidenced by esophago-gastro-duodenoscopy (EGD) with biopsy and Esophageal Impedance Monitoring (EIM)
  Interventions: Procedure: Esophago-gastro-duodenoscopy (EGD) with biopsy; Procedure: Esophageal Impedance Monitoring (EIM)
- Control: CC/GER- presence of chronic cough and absence of GER by esophago-gastro-duodenoscopy (EGD) with biopsy and Esophageal Impedance Monitoring (EIM)
  Interventions: Procedure: Esophago-gastro-duodenoscopy (EGD) with biopsy; Procedure: Esophageal Impedance Monitoring (EIM)

INTERVENTIONS:
Procedure: Esophago-gastro-duodenoscopy (EGD) with biopsy
Procedure: Esophageal Impedance Monitoring (EIM)

SUMMARY:
Using an active cohort of children in whom Airway and gastrointestinal endoscopy will be performed, investigators will conduct a chart review to obtain relevant clinical data and the investigators will use an aliquot of airway sample obtained during the clinically indicated bronchoscopy for microbiome analysis. A case-control study design will be used to study whether subjects with CC with GER have a distinct lung microbiome and increased inflammation as compared with subjects with CC without GER and to determine whether the microbiome and degree of inflammation is related to the type of GER (acidic versus nonacidic).

ELIGIBILITY:
Inclusion Criteria:

* Children (Age 0 - 24 years) referred to the NYU Pediatric AeroDigestive Center to evaluate for CC (>4weeks).

Exclusion Criteria:

* Antibiotic or steroids (inhaled or systemic) use within the prior one-week. Rationale: Antibacterial drugs and immune-modulators are confounders that may impact the microbiome and inflammation. While longer period free of Antibacterial drugs and immune-modulators would be desired, it would be unethical and it is not the usual standard of care to withdraw treatment for longer periods of time.
* Interstitial Lung Disease or pneumonia on X-ray
* Cystic fibrosis
* Primary ciliary dyskinesia
* Immunodeficiency syndromes
* Major airway abnormalities
* Proton pump inhibitor/H2-receptor antagonist therapy within the prior 2 weeks

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (Age 0 - 24 years) referred to the NYU Pediatric AeroDigestive Center to evaluate for CC (>4weeks).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Reflux Finding Score (RFS) in CC/GER- group and CC/GER+ group | 2 Years
Comparison of bronchoscopic secretions scoring system (BSSS) in CC/GER- group and CC/GER+ group | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail N Kazachkov, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States